CLINICAL TRIAL: NCT01148004
Title: The Influence of Ritonavir, Alone and in Combination With Lopinavir, on Fenofibric Acid Pharmacokinetics in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 100124; 10-CC-0124
Record Dates: First submitted 2010-06-18; First posted 2010-06-22 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2013-07-29

CONDITIONS: HIV; Fenofibrate; Protease Inhibitors; Hypertriglyceridemia; Glucuronosyltransferase
Keywords: HIV; Hypertriglyceridemia; Protease Inhibitors; Healthy Volunteer; HV
MeSH Terms: conditions — Hypertriglyceridemia | interventions — Fenofibrate; Ritonavir; Lopinavir

INTERVENTIONS:
Drug: Fenofibrate
Drug: Ritonavir
Drug: Lopinavir/Ritonavir

SUMMARY:
Background:

- Patients infected with the human immunodeficiency virus (HIV) are often treated with protease inhibitors that help fight HIV infection. However, these medications often increase blood cholesterol levels, particularly triglycerides and low-density lipoproteins, and can lead to heart disease and other problems. Patients may take drugs known as fibrates (such as gemfibrozil (Lopid )) to lower triglyceride levels, but even with maximum approved doses patients often cannot reach goal triglyceride levels. Research suggests that fibrates and certain HIV medications, such as ritonavir and lopinavir/ritonavir, may interact and decrease the effectiveness of the fibrate treatment. More research is needed to determine the best drug to lower triglyceride levels in HIV patients who are receiving protease inhibitor therapy.

Objectives:

- To evaluate the drug-drug interaction between fenofibrate and protease inhibitors lopinavir/ritonavir and ritonavir.

Eligibility:

- Healthy individuals between 18 and 60 years of age.

Design:

* This study will require a screening visit and 18 study visits. The screening visit will take 3 to 4 hours, and can occur 7 to 30 days before starting the study. The rest of the study, not including the screening visit, is 48 days. Three of the visits will take about 12 hours, and the remaining 15 visits will take about 1 hour.
* For study days 1 to 7, participants will take fenofibrate alone. Participants will keep a daily record of medication doses and any side effects.
* For study days 8 to 27, participants will take fenofibrate and ritonavir. Participants will keep a daily record of medication doses and any side effects.
* For study days 29 to 48, participants will take fenofibrate and lopinavir/ritonavir. Participants will keep a daily record of medication doses and any side effects.
* Participants will have regular study visits to provide blood samples for research and monitoring.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has enhanced the life expectancy of human immunodeficiency virus (HIV) infected patients, making HIV a manageable chronic disease for many patients. Patients with HIV are prone to lipid abnormalities secondary to HIV infection and antiretroviral therapy, particularly HIV protease inhibitors (PI). PI containing regimens that contain boosting doses of ritonavir (RTV) (i.e., 100 200 mg once or twice daily) often cause significant increases in total cholesterol, low density lipoprotein cholesterol, and triglycerides. Therapy for isolated hypertriglyceridemia includes fibric acid derivatives, such as gemfibrozil (GFZ) or fenofibrate; however, despite treatment with these agents, triglyceride levels often remain elevated in HIV infected patients treated with HAART. Many factors likely contribute to the incomplete effectiveness of fibrates in these patients. One possible contributing factor may be a clinically significant interaction between HAART and fibrates. We recently reported a mean 41 percent decrease in GFZ area under the curve when administered with the PI combination lopinavir/ritonavir (LPV/r). To determine whether a similar interaction exists with fenofibrate, this study will characterize the impact of RTV and LPV/r on the pharmacokinetic (PK) profile of fenofibrate (Tricor formulation), after a single 145 mg oral dose, administered to healthy volunteers. In a single sequence study design, 13 subjects will receive a single 145 mg dose of fenofibrate on three occasions: before and after 14 days of RTV 100 mg twice daily, and after 14 days of LPV/r 400/100 mg twice daily. With the exclusion of the screening period, the total duration of the study will be 48 days. Fenofibric acid (FFA) PK will be determined for all 3 sampling periods and compared. Results from this study will inform us about a potentially clinically relevant drug drug interaction between fenofibrate and RTV boosted PI combinations. This information may therefore assist clinicians in choosing triglyceride lowering therapy for their HIV infected patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

A subject will be considered eligible for this study only if all of the following criteria are met:

* Between the ages of 18 and 60 years
* Healthy according to medical history and physical examination
* Laboratory values: normal liver function tests (ALT less than or equal to 41 units/L, AST less than or equal to 34 units/L, total bilirubin less than or equal to 1.0 mg/dL, and direct bilirubin less than or equal to 0.2 mg/dL); serum creatinine less than or equal to ULN; hemoglobin greater than or equal to 12 g/dL (for both males and females)

  a. For patients with a history of Gilbert's Syndrome, patients with a total bilirubin that is greater than 1.0 mg/dL will be considered eligible for study participation if direct bilirubin is within normal limits (direct bilirubin < 0.2 mg/dL)
* Normal ECG with no history of cardiac arrhythmias or conduction abnormalities
* Females of child bearing potential who are able and willing to prevent pregnancy by

  * a. practicing abstinence or
  * b. using non hormonal effective methods of birth control, such as condoms or

diaphragms during the study period and for 1 month after study completion

EXCLUSION CRITERIA:

A subject will be ineligible for this study if 1 or more of the following criteria are met:

* Concomitant routine therapy with any prescription, over the counter, herbal, or holistic medications, including hormonal contraceptives by any route and any investigational drugs for 30 days prior to study participation

  * Concomitant therapy (chronic or intermittent) with any prescription, over the counter, or herbal drugs will not be allowed during the study duration
  * Intermittent use of acetaminophen, non-steroidal anti-inflammatory medications (i.e., ibuprofen), and loperamide will be allowed to be taken according to each manufacturer s recommendations during the study, but will not be allowed on the days of PK blood sampling
  * A daily multivitamin with minerals will be allowed during the study, according to the subject s wishes
* Inability to obtain venous access for blood sample collection
* The presence or history of any of the following:

  * Diabetes mellitus (clinical diagnosis based on current guidelines)
  * HIV infection
  * Pulmonary disease (e.g. uncontrolled asthma, chronic obstructive pulmonary disease, etc.)
  * Cardiac disease (e.g. heart failure, history of arrhythmia, or abnormal ECG results during screening, etc.)
  * Hypertension (systolic blood pressure greater than 145 mmHG or diastolic blood pressure greater than 90 mmHg)
  * Renal disease (chronic or acute renal failure or insufficiency)
  * Hepatitis (as assessed by patient interview) or hepatic impairment
  * Pancreatitis
  * Bleeding disorders (e.g. hemophilia, gastrointestinal or intracranial bleeding)
  * Organ transplant
  * Seizure disorders, with the exception of childhood febrile seizures in the past
  * Schizophrenia or other psychiatric illnesses that may interfere with the subject s ability to participate in the study
  * Any condition that may interfere with the interpretation of the study results or not be in the best interest of the subject in the opinion of the investigators
* Positive serum or urine pregnancy test or breastfeeding female
* The presence of persistent diarrhea or malabsorption that would interfere with the subject s ability to absorb drugs
* Drug or alcohol abuse that may impair safety or adherence
* History of intolerance or allergic reaction to LPV/r, RTV, or fenofibrate
* Fasting total cholesterol greater than 240 mg/dL or fasting triglycerides greater than 400 mg/dL
* Fasting glucose greater than 100 mg/dL
* Use of tobacco products, including cigarettes and chewing tobacco

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-05-13; Primary Completion 2013-07-29 (Actual); Study Completion 2013-07-29 (Actual)

PRIMARY OUTCOMES:
Fenofibratae pharmacokinetic parameter values | 48 days from study day 1 (after screening has been completed)

CONTACTS AND LOCATIONS:
Overall Officials: Scott R Penzak, Pharm.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Penzak SR, Chuck SK. Management of protease inhibitor-associated hyperlipidemia. Am J Cardiovasc Drugs. 2002;2(2):91-106. doi: 10.2165/00129784-200202020-00003. PMID 14727985
- [Background] Grunfeld C, Tien P. Difficulties in understanding the metabolic complications of acquired immune deficiency syndrome. Clin Infect Dis. 2003;37 Suppl 2:S43-6. doi: 10.1086/375886. PMID 12942373
- [Background] Sax PE. Strategies for management and treatment of dyslipidemia in HIV/AIDS. AIDS Care. 2006 Feb;18(2):149-57. doi: 10.1080/09540120500161843. PMID 16338773